CLINICAL TRIAL: NCT01222078
Title: Evaluation of the Safety and Tolerability of Re-dosing With Intravenous (iv) Otelixizumab in Adult Subjects With Newly Diagnosed Type 1 Diabetes Mellitus
Brief Title: Investigating Re-Dosing With Otelixizumab in Adults With Newly-Diagnosed Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A Phase 3 study recently reported and demonstrated that the dose of otelixizumab in OTX113390 is not effective.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113390; 2010-019157-17 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-18 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: newly diagnosed type 1 diabetes mellitus; re-treatment; intravenous otelixizumab; beta-cell preservation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — otelixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- otelixizumab (Experimental): otelixizumab
  Interventions: Biological: otelixizumab

INTERVENTIONS:
Biological: otelixizumab — Two treatment courses of otelixizumab given 6 months apart. Each treatment course will consist of 8 consecutive days of otelixizumab intravenous infusions (each given over 30 minutes).

SUMMARY:
The purpose of this study to assess the safety and tolerability of re-dosing at 6 months with otelixizumab (given as an 8-day series of intravenous infusions) in adult subjects with newly diagnosed type 1 diabetes mellitus

DETAILED DESCRIPTION:
The primary objective of this phase IIa, open-label, multi-centre study is to assess the safety, tolerability and immunogenicity of re-dosing at 6 months with an 8 consecutive day series of otelixizumab intravenous (IV) infusions in 8 adult subjects with newly diagnosed type 1 diabetes mellitus (T1DM). Although it is hoped that the β cell preserving effect of otelixizumab will be long-lasting, it is possible that the effect may decline over time and thus T1DM subjects may require re-treatment. Six months is the minimum time expected between treatments.

After baseline assessments, eligible subjects will receive 8 consecutive days of otelixizumab infusions, each given over a 30 minute period. Prophylaxis for cytokine release syndrome AEs will be given. At Month 6, following a review of any new medical conditions, concomitant medications, lymphocyte count, Epstein Barr Virus (EBV) viral load and other re-dosing eligibility criteria, subjects will be re-treated with the same dosing regimen. Subjects will be followed for 24 months in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 45 years. Women are allowed if they are of non-childbearing potential or agree to use one of the contraception methods listed in the protocol.
* Diagnosis of type 1 autoimmune diabetes mellitus according to ADA and WHO criteria
* No more than 90 days between diagnosis and the first dose of study drug.
* Currently requires insulin for T1DM treatment, or has required insulin at some time between diagnosis and the first dose of study drug.
* Positive for one or more of the autoantibodies typically associated with T1DM: antibody to glutamic acid decarboxylase (anti-GAD); antibody to protein tyrosine phosphatase-like protein (anti-IA-2); or insulin autoantibodies (IAA). A subject who is positive for insulin autoantibodies (IAA) and negative for the other autoantibodies will only be eligible if the subject has used insulin for less than 7 days total.
* Stimulated C-peptide level greater than 0.20 nmol/L and less than or equal to 3.50 nmol/L
* Body mass index not greater than 32 kg/m2.
* QTc <450 millisecond (msec) or <480msec for patients with Bundle Branch Block

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant from the beginning of the screening period or at least 14 days prior to initial dosing until at least 60 days after the last dose of the second treatment course of study drug.
* Current or prior malignancy, other than non-melanoma skin cancer (subject must have had fewer than 5 occurrences of non-melanoma skin cancer, and the last occurrence must not be within 3 months of study entry).
* Clinically significant abnormal laboratory values during the Screening period, other than those due to T1DM. Permitted ranges for selected laboratory values are shown in the protocol. A clinically significant abnormal value will not result in exclusion if, upon re test, the abnormality is resolved or becomes clinically insignificant.
* Significant and/or active disease in any body system likely to increase the risk to the subject or interfere with the subject's participation in or completion of the study. Examples of significant diseases include, but are not limited to, coronary artery disease, congestive heart failure, uncontrolled hypertension, renal failure, emphysema, history of bleeding peptic ulcers, history of seizure(s), addiction to illicit drugs, and alcohol abuse.
* Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), presence of hepatitis B surface antigen (HBsAg), positive hepatitis C test result within 3 months of screening
* Significant systemic infection during the 6 weeks before the first dose of study drug (e.g., infection requiring hospitalisation, major surgery, or IV antibiotics to resolve; other infections, e.g., bronchitis, sinusitis, localised cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-by-case basis by the investigator regarding whether they are serious enough to warrant exclusion).
* History of current or past active tuberculosis infection and or latent tuberculosis infection. Further details are given in the protocol.
* A positive test for human immunodeficiency virus (HIV) antibody or risk factors which predispose subject to HIV infection.
* EBV viral load greater than or = to 10,000 copies per 10xe6 peripheral blood mononuclear cells (PBMCs) as determined by quantitative polymerase chain reaction (qPCR). If there is any clinical suspicion that a subject who is EBV seronegative and with EBV PCR <10,000 copies per 10xe6 PBMCs has symptoms consistent with infectious mononucleosis prior to administration of study drug, then a monospot test result must be negative before the subject can be dosed.
* A positive test for syphilis.
* Had a potent immunosuppressive agent (e.g., systemic high-dose corticosteroids on a chronic basis, methotrexate, cyclosporine, or anti-TNF agents) within the 30 days before the first dose of study drug, or expecting to require such treatment within 3 months after the last dose of study drug. (Intranasal, inhaled, and topical corticosteroid medications are permitted if used at recommended dosages.)
* Used an atypical antipsychotic drug (e.g., risperidone [Risperdal], quetiapine [Seroquel], or clozapine [Clozaril]) within the 30 days before first dose of study drug, or expecting to require such treatment during the study.
* Received a vaccine within the 30 days before the first dose of study drug, or expecting to require a vaccine during the dosing period or the 30 days after the last dose of study drug.
* Previously received otelixizumab or any other anti CD3 monoclonal antibody, e.g., OKT3 (muromonab or Orthoclone), ChAglyCD3, or hOKT3γ1 (ala ala), or not willing to refrain from using any such antibody for the planned duration of study participation (18 months after the last dose of study drug).
* Previously received an anti lymphocyte monoclonal antibody, such as anti-CD20, anti-thymocyte globulin (ATG), rituximab (Rituxan), or alemtuzumab (Campath), or planning to use any such antibody during the planned duration of study participation (18 months after the last dose of study drug).
* Had an investigational drug within the 3 months before the first dose of study drug or planning to take an investigational drug within18 months of the last dose of study drug.
* Have donated any plasma or blood within 45 days before the first dose of study drug.
* Prior allergic reaction, including anaphylaxis, to any human, humanised, chimeric, or rodent antibody.
* Undergone a major surgical procedure within 30 days before the first dose of study drug, or planning to undergo any such surgery within 3 months after the last dose of study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2011-05-19 (Actual); Study Completion 2011-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Paris, France
- GSK Investigational Site, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing the attached study results summary with a conclusion.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one site in France during the period 22 November 2010 to 19 May 2011 and was planned to enroll 8 participants. But only one participant was enrolled and received a single course of study medication. No participants were re-dosed.
Groups:
- Otelixizumab: Participant received a single dose of otelixizumab intravenous (IV) infusions each given over a 30 minute period on 8 consecutive days in order: 0.1 milligrams (mg), 0.2 mg, 0.3 mg, 0.5 mg, 0.5 mg, 0.5 mg, 0.5 mg, 0.5 mg thus total dose 3.1 mg. Participant received prophylactic oral ibuprofen 400-800 mg 2 hours before start of infusion (SOI), 2 hours after SOI, 6 hours after SOI and at bedtime. Participant received 5-10 mg oral levocetirizine 1 hour prior to each infusion. Participant was about to receive same study drug dosing after 6 months, though not received.
Period: Overall Study
Arm/Group | Otelixizumab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Early termination of the study | 1

BASELINE CHARACTERISTICS:
Groups:
- Otelixizumab: Participant received a single dose of otelixizumab IV infusions each given over a 30 minute period on 8 consecutive days in order: 0.1mg, 0.2 mg, 0.3 mg, 0.5 mg, 0.5 mg, 0.5 mg, 0.5 mg, 0.5 mg thus total dose 3.1 mg. Participant received prophylactic oral ibuprofen 400-800 mg 2 hours before SOI, 2 hours after SOI, 6 hours after SOI and at bedtime. Participant received 5-10 mg oral levocetirizine 1 hour prior to each infusion. Participant was about to receive same study drug dosing after 6 months, though not received.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (NA) — Only one participant enrolled
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious AEs (SAEs)
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Study was early terminated and participant withdrew on study Day 164.
Time Frame: Up to Month 24
Population: Safety Population consisted of participants who had received at least one dose of infusion.
Measure: Number; unit: Participants
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Participants
  Any AEs | 1
  Any SAEs | 0

2. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was assessed at sitting position at Baseline and 1 to 7 hours of post-infusion of first treatment period. Day 1 value was considered to be Baseline value. Change from Baseline was planned to be calculated as any post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

3. Primary Outcome: Mean Change From Baseline in Respiration Rate
Description: Respiration rate was assessed at sitting position at Baseline and post-treatment. Day 1 value was considered to be Baseline value. Change from Baseline was planned to be calculated as any post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

4. Primary Outcome: Mean Change From Baseline in Temperature
Description: Temperature was recorded at sitting position at Baseline and post treatment. Day 1 value was considered to be Baseline value. Change from Baseline was planned to be calculated as any post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

5. Primary Outcome: Mean Change From Baseline in Heart Rate
Description: Heart rate was recorded at sitting position at Baseline and post-treatment period. Day 1 value was considered to be Baseline value. Change from Baseline was planned to be calculated as any post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

6. Primary Outcome: Number of Participants With Values Outside the Normal Range for Vitals
Description: Vital included assessment of SBP, DBP, respiration rate, heart rate and temperature were assessed at sitting position. Participant did not received re-dose of second treatment period and withdrew on study Day 164 because of early study termination.
Time Frame: Up to Month 24
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Participants
  SBP and DBP | 1
  Respiration rate | 1
  Heart rate | 1
  Temperature | 0

7. Primary Outcome: Mean Change From Baseline in Value of Albumin and Total Protein
Description: Clinical chemistry parameters were planned to be analyzed from Baseline to Month 24. Day 1 value was considered to be Baseline value. Change from Baseline was planned to be calculated as any post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

8. Primary Outcome: Mean Change From Baseline in Value of Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatinine Kinase, Follicle Stimulating Hormone, Gamma Glutamyl Tranferase and Lactate Dehydrogenase
Description: as for outcome 7
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

9. Primary Outcome: Mean Change From Baseline in Value of Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid
Description: as for outcome 7
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

10. Primary Outcome: Mean Change From Baseline in Value of Calcium, Chloride, Carbon Dioxide Content/Bicarbonate, Glucose, Potassium, Magnesium, Sodium, Inorganic Phosphorus and Urea/Blood Urea Nitrogen
Description: as for outcome 7
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

11. Primary Outcome: Mean Change From Baseline in Value of Estradiol
Description: as for outcome 7
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

12. Primary Outcome: Mean Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count and White Blood Cell Count
Description: Hematology parameters were planned to be analyzed from Baseline to Month 24. Day 1 value was considered to be Baseline value. Change from Baseline was planned to be calculated as any post-Baseline value minus Baseline value.
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

13. Primary Outcome: Mean Change From Baseline in Glycosylated Hemoglobin Value
Description: as for outcome 12
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

14. Primary Outcome: Mean Change From Baseline in Hemoglobin Value
Description: as for outcome 12
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

15. Primary Outcome: Mean Change From Baseline in Red Blood Cell Count
Description: as for outcome 12
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

16. Primary Outcome: Mean Epstein-Barr Virus (EBV) Viral Load
Description: Levels of EBV were assessed periodically using Quantitative Polymerase Chain Reaction. If a participant had an EBV viral load of >=10,000 copies per 10^6 Peripheral Blood Mononuclear Cells (PBMCs) at any visit, the test was repeated as soon as possible to confirm this result. If the result was confirmed, the test was repeated weekly for 2 weeks or until the count decreases to < 10,000 copies per 10^6 PBMCs, whichever was longer. The EBV Load remained zero throughout the study. Participant did not received re-dose of second treatment period and withdrew on study Day 164 because of early study termination. The viral load was to measure using unit copies per 10^6 Peripheral Blood Mononuclear Cells (PBMCs)
Time Frame: Up to Month 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Copies per 10^6 PBMCs
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Copies per 10^6 PBMCs | 0 (NA) — The value remained zero throughout the study

17. Primary Outcome: Mean Change in Total Lymphocyte Count
Description: Total lymphocyte count was planned to be analyzed up to Month 24.
Time Frame: Baseline and up to Month 24
Population: Safety Population. Because of the early termination of the study this endpoint was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

18. Primary Outcome: Mean Change in CD4+ and CD8+ T-cell Counts
Description: CD4+ and CD8+ T cells were planned to be measured before, during and after dose 1, 4 and 8 of first treatment course. Because of the early termination of the study the data was not analyzed.
Time Frame: Days 1, 4 and 8 of each treatment course
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent total lymphocytes
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Percent total lymphocytes | NA (NA) — As study was early terminated, data was not analyzed

19. Primary Outcome: Mean Change in Circulating Peripheral T Lymphocytes
Description: Circulating peripheral T lymphocytes were planned to be measured before, during and after dose 1, 4 and 8 of first treatment course. Because of the early termination of the study the data was not analyzed.
Time Frame: Days 1, 4 and 8 of each treatment course
Population: Safety Population
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
GI/L | NA (NA) — As study was early terminated, data was not analyzed.

20. Primary Outcome: Mean Change in Circulating Peripheral CD4+ and CD8+ Subset Counts
Description: Circulating peripheral CD4+ and CD8+ T cells were planned to be measured before, during and after dose 1, 4 and 8 of first treatment course. Because of the early termination of the study the data was not analyzed.
Time Frame: Days 1, 4 and 8 of each treatment course
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent total lymphocytes
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Percent total lymphocytes | NA (NA) — As study was early terminated, data was not analyzed

21. Primary Outcome: Mean Serum Levels of Anti-otelixizumab Binding Antibodies
Description: Antibodies to otelixizumab were planned to be measured at Baseline and at specified post-Baseline visits using a validated immunoassay. If a positive result was detected, the samples were analyzed further in a neutralizing antibody assay to determine if the antibodies were neutralizing. The 12 and 24 month samples were only be taken if a participant had a positive result for antibodies at the last tested time point (Month 9) or if the Month 9 test results were not available.
Time Frame: Up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

22. Primary Outcome: Proportion of Anti-otelixizumab Neutralizing Antibodies
Description: as for outcome 21
Time Frame: Up to Month 24
Population: Safety Population. Because of the early termination of the study the data was not collected.
Arm/Group | Otelixizumab
Number analyzed (Participants) | 0

23. Secondary Outcome: Mean Circulating Peripheral T Lymphocytes Count
Description: as for outcome 19
Time Frame: Day 1, 4 and 8 of each treatment course
Population: Safety Population
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
GI/L | NA (NA) — As study was early terminated, data was not analyzed

24. Secondary Outcome: Mean Circulating CD4+ and CD8+ Subset Counts
Description: as for outcome 20
Time Frame: Days 1, 4 and 8 of each treatment course
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent total lymphocytes
Groups:
- Overall Study Arm: Participant received a single dose of otelixizumab IV infusions each given over a 30 minute period on 8 consecutive days in order: 0.1mg, 0.2 mg, 0.3 mg, 0.5 mg, 0.5 mg, 0.5 mg, 0.5 mg, 0.5 mg thus total dose 3.1 mg. Participant received prophylactic oral ibuprofen 400-800 mg 2 hours before SOI, 2 hours after SOI, 6 hours after SOI and at bedtime. Participant received 5-10 mg oral levocetirizine 1 hour prior to each infusion. Participant was about to receive same study drug dosing after 6 months, though not received.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 1
Percent total lymphocytes | NA (NA) — As study was early terminated, data was not analyzed

25. Secondary Outcome: Mean Saturation of CD3 Antigen on Peripheral Blood T Cells
Description: Assessment of CD3 antigen was planned to be done on Day 1, 4 and 8 of first treatment course. The data was planned to be presented with unit Molecules of Equivalent Soluble Fluorochrome (MESF). Because of the early termination of the study the data was not analyzed.
Time Frame: Days 1, 4 and 8 of each treatment course
Population: Safety Population
Measure: Mean (Standard Deviation); unit: MESF
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
MESF | NA (NA) — As study was early terminated, data was not analyzed

26. Secondary Outcome: Mean Individual Serum Concentrations of Otelixizumab
Description: Because of the early termination of the study the data was not analyzed.
Time Frame: Pre-dose and EOI on Dosing Day 1, EOI on Dosing Days 2, 3, 5-7 and Pre-dose, EOI, 6 hours post SOI on Dosing days 4 and 8 of each treatment course
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Nanograms per milliliter (ng/mL) | NA (NA) — As study was early terminated, data was not analyzed

27. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Otelixizumab
Description: Because of the early termination of the study the data was not analyzed.
Time Frame: as for outcome 26
Population: Safety Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
ng/mL | NA (NA) — As study was early terminated, data was not analyzed

28. Secondary Outcome: Time to Cmax (Tmax) of Otelixizumab
Description: Because of the early termination of the study the data was not analyzed.
Time Frame: as for outcome 26
Population: Safety Population
Measure: Median (Full Range); unit: hours
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
hours | NA [NA to NA] — Value could not be determined due to insufficient quantifiable concentrations and the study was early terminated.

29. Secondary Outcome: Area Under the Serum Concentration-time Curve [AUC(0-tlast)] of Otelixizumab
Description: Because of the early termination of the study the data was not analyzed.
Time Frame: as for outcome 26
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Hours times nanograms per milliliter
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
Hours times nanograms per milliliter | NA (NA) — Value could not be determined due to insufficient quantifiable concentrations and the study was early terminated.

30. Secondary Outcome: Time of Last Observed Quantifiable Concentration (Tlast) of Otelixizumab
Description: Because of the early termination of the study the data was not analyzed.
Time Frame: as for outcome 26
Population: Safety Population
Measure: Median (Full Range); unit: hours
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
hours | NA [NA to NA] — Value could not be determined due to insufficient quantifiable concentrations and the study was early terminated.

31. Secondary Outcome: Terminal Phase Half-life (Thalf) of Otelixizumab
Description: Because of the early termination of the study the data was not analyzed.
Time Frame: as for outcome 26
Population: Safety Population
Measure: Median (Full Range); unit: hours
Arm/Group | Otelixizumab
Number analyzed (Participants) | 1
hours | NA [NA to NA] — Value could not be determined due to insufficient quantifiable concentrations and the study was early terminated.

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were reported since first dose of investigational product up to Month 24.
Description: Safety Population consisted of participants who had received at least one dose of infusion.
Arm/Group | Otelixizumab
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Otelixizumab (N=1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.